CLINICAL TRIAL: NCT05280145
Title: Assessment of the echOpen Ultra-portable Ultrasound Device in Daily Use by Clinicians. Part II: Detection of Pyelocaliceal Dilation and Hepatic Steatosis
Brief Title: Efficacy of the echOpen Device to Detect Pyelocaliceal Dilation and Hepatic Steatosis
Acronym: CLIN-ECHO-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ECHOPEN (Industry); EIT Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP211147; 2021-A02168-33 (Other: IDRCB)
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hepatic Steatosis; Fatty Liver; Hydronephrosis
Keywords: Ultrasound; Ultrasonography; Point-of-care-ultrasound; Hepatic Steatosis; pyelocaliceal system
MeSH Terms: conditions — Fatty Liver; Hydronephrosis

STUDY DESIGN:
Intervention Model Description: A single group, comparative, non-randomized, controlled study. Each patient represents her/his own control: the patient is examined consecutively with the echOpen probe, then with the probe routinely used in the department
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients benefitting ultrasound examination (Experimental): This is the only arm of the study. Patients with an indicative clinical picture that leads the clinician to resort to the use of an ultrasound to potentially support the diagnosis, will be examined depending on clinical presentation for either the presence of pyelocaliceal dilatation, or hepatic steatosis. The patients will be assessed first with the echOpen device and second witn an ultrasound routinely used in the department. In a case of discordance between the assessments made with echOpen and the usual ultrasound device, an independent referent radiologist will use a standard ultrasound machine to constitute the gold standard (GS) rating. If the latter is not available to carry out the third ultrasound scan within a timeframe deemed clinically acceptable, then the evaluation will be carried out in a delayed manner, using the video loops and image captures saved during the two initial ultrasound scans.
  Interventions: Device: EchOpen ultra-portable ultrasound device; Device: Ultrasound device routinely used in the department; Procedure: Ultrasound examination by an independent referent radiologist

INTERVENTIONS:
Device: EchOpen ultra-portable ultrasound device — Depending on the clinical picture, the patient is examined with EchOpen to detect the presence or absence of pyelocaliceal dilatation or hepatic steatosis
Device: Ultrasound device routinely used in the department — Patient who was first examined with EchOpen, is secondarily examined with an ultrasound probe used routinely in the department to detect pyelocaliceal dilatation or hepatic steatosis
Procedure: Ultrasound examination by an independent referent radiologist — In a case of discordance between the assessments made with echOpen and the usual ultrasound device, an independent referent radiologist will use a standard ultrasound machine to constitute the gold standard (GS) rating. If the latter is not available to carry out the third ultrasound scan within a timeframe deemed clinically acceptable, then the evaluation will be carried out in a delayed manner, using the video loops and image captures saved during the two initial ultrasound scans.

SUMMARY:
In recent years, portable and ultra-portable ultrasound devices are increasingly used by the non radiologists, notably cardiologists or obstetrician gynecologist, at the patient's bedside to visualize and measure anatomical structures and fluid and provide the clinical examination with additional signs allowing quicker and more confident clinical decisions.

This innovative approach is slowed down by the accessibility of these miniaturized devices, the price of which remains high.

The echOpen device includes an ultra-portable ultrasound probe and a mobile application that allows the image to be displayed on a smartphone via a WIFI protocol.

The objective of the clinical investigation is to show that the echOpen device, using three frequencies 3.5 Mhz, 5.0 Mhz and 7.5 Mhz, allows identifying the semiological signs or anatomical structures of interest located at several depths of the body, with a performance similar to other devices routinely used in clinical departments.

DETAILED DESCRIPTION:
The echOpen device includes an ultrasound probe and a mobile application. The mechanical probe emits at three ultrasound frequencies, 3.5 Mhz, 5.0 Mhz and 7.5 Mhz, which allows the exploration of the interior of the body at different depths in a non-invasive and non-irradiating manner.

Thus, the purpose of the echOpen device is, on one hand, to guide the diagnosis during the clinical examination and, on the other hand, to identify anatomical structures in order to assist in management.

The objective of the clinical investigation is to demonstrate that the echOpen device is able to identify semiological signs and localize anatomical structures at different depths of the body, with a performance not inferior to that of other ultrasound devices, routinely employed in hospital clinical departments.

The signs of interest (i.e. detection of pyelocaliceal dilation (3.5 Mhz) and hepatic steatosis (5.0 Mhz) were chosen for their clinical usefulness (their identification during the clinical examination constitutes an argument for orientation and/or severity) and for their prevalence in the study population.

An ultrasound probe in use in the hospital clinical departments where the investigation takes place will be employed as a comparator to judge the performance of the echOpen device.

This clinical investigation is part of a CE marking procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years old)
* Patient having signed the informed consent to participate in this clinical investigation
* Patient affiliated to the social security scheme
* Patient arriving in the hospital clinical ward (own initiative or by emergency services) whose clinical symptomatology suggests the presence of pathological elements which would be visible using an ultrasound probe in the following cases:

  * Search for pyelocaliceal dilation: patient consulting for abdominal and/or lumbar pain and/or iliac fossa, fever, pain in the right or left iliac fossa, anuresis
  * Search for hepatic steatosis: in a case of global clinical examination, abnormal laboratory test results, known or suspected metabolic disease, any situation suggesting the presence of hepatic steatosis

Exclusion Criteria:

* Minor patient (age < 18 years)
* Patients under the State Medical Assistance (AME)
* Obese patient (body mass index > 29.9)
* Patient in too serious condition for the clinical examination to be done fully and/or with additional exploratory time
* Unstable patient: need for immediate care, impossibility to carry out a thorough clinical examination including interview, palpation, auscultation, percussion
* Known allergy to ultrasound gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-08-21 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Presence of Pyelocaliceal dilation | Day 0
  Pyelocaliceal system assessment by using echOpen or a portable ultrasound routinely used in the department and scored as follows: 0, normal condition; 1, normal parenchyma, dilated renal pelvis, undilated calyces; 2, normal parenchyma, renal pelvis and calyces dilated, papillary impression preserved; 3, parenchyma thinned, significant pyelocaliceal dilation with bulging calyxes and disappearance of the papillary impression; 4, very thinned parenchyma, massive pyelocaliceal dilation, disappearance of the pyelocaliceal differentiation.
Presence of Hepatic steatosis | Day 0
  Hepatic steatosis assessment by using echOpen or a portable ultrasound routinely used in the department and scored on the base of liver echogenicity as follows: 0, normal condition; 1, local hyperechogenicity; 2, diffuse hyperechogenicity

SECONDARY OUTCOMES:
Pyelocaliceal dilation determined using a gold standard procedure | Day 0
  Pyelocaliceal system assessment by by an independent referent radiologist using a standard ultrasound machine and scored as follows: 0, normal condition; 1, normal parenchyma, dilated renal pelvis, undilated calyces; 2, normal parenchyma, renal pelvis and calyces dilated, papillary impression preserved; 3, parenchyma thinned, significant pyelocaliceal dilation with bulging calyxes and disappearance of the papillary impression; 4, very thinned parenchyma, massive pyelocaliceal dilation, disappearance of the pyelocaliceal differentiation.
Hepatic steatosis determined using a gold standard procedure | Day 0
  Hepatic steatosis assessment by by an independent referent radiologist using a standard ultrasound machine and scored on the base of liver echogenicity as follows: 0, normal condition; 1, local hyperechogenicity; 2, diffuse hyperechogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme BOKOBZA, MD, Principal Investigator — AP-HP, Cochin Hospital
Locations (4):
- France (4):
  - Avicenne Hospital - APHP- Hepatology Department, Bobigny
  - Groupe Hospitalier Sud Ile de France (GHSIF) - Emergency Department, Melun
  - APHP COCHIN HOSPITAL - Emergency Department, Paris
  - Paul Brousse Hospital - APHP - Hepatobiliary Center, Villejuif